CLINICAL TRIAL: NCT03715543
Title: Surgical Resection of the Greater Splanchnic Nerve in Subjects Having Heart Failure With Preserved Ejection Fraction: First-in-human Feasibility Trial
Brief Title: Surgical Resection of the Greater Splanchnic Nerve in Subjects Having Heart Failure With Preserved Ejection Fraction
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Noblewell (Industry)
Collaborators: Coridea (Industry); Axon Therapies (Unknown)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: GSN FIH Study
Record Dates: First submitted 2018-08-16; First posted 2018-10-23 (Actual); Last update posted 2020-06-30 (Actual); Status verified 2020-06

CONDITIONS: Heart Failure With Preserved Ejection Fraction

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Surgical Resection Arm (Experimental): Surgical Resection of the Greater Splanchnic Nerve
  Interventions: Procedure: Surgical Resection of the Greater Splanchnic Nerve

INTERVENTIONS:
Procedure: Surgical Resection of the Greater Splanchnic Nerve — Video-Assisted Thoracoscopic Surgery (VATS) is performed under general anesthesia using existing, CE marked instrumentation. Two or more 5 mm incisions are used to pass a tiny video camera and a single dissecting instrument into the chest. These small ports are advantageous because the chance for infection and wound dehiscence are drastically reduced. This allows for a faster recovery by the patient and a greater chance for the wound to heal.
  In the procedure the GSN will be identified visually or through stimulation-induced hemodynamic reflex. The GSN will then be ablated using standard techniques. If there are multiple branches of the GSN, each branch will be systematically identified and ablated.

SUMMARY:
We believe that blocking of the Greater Splanchnic Nerve (GSN) will stop Sympathetic Nervous System (SNS) activity from reaching the splanchnic vessels and result in a redistribution of blood volume back into the splanchnic reservoir, which will result in reduction of central venous, pulmonary and right and left heart pressures. For patients having Heart Failure With Preserved Ejection Fraction (HFpEF) we expect these changes to improve dyspnea and capacity to exercise, improve quality of life, increased diuretic responsiveness, Furthermore, the expected benefits of unloading the central venous and arterial system through GSN ablation should improve hemodynamic control and lessen the incidence and severity of acute decompensations leading to reduced re-hospitalizations and associated healthcare costs. This has the potential for significant social and healthcare impact.

DETAILED DESCRIPTION:
Heart failure (HF) is a major and growing public health problem with more than 5 million identified cases and an incidence of over 600,000 new cases per year in the United States alone. Close to 1 million hospitalizations for heart failure occur annually, accounting for over 6.5 million hospital days and a substantial portion of the estimated $37.2 billion that is spent each year on HF in the United States. Nearly half of all patients with HF have so called heart failure with preserved ejection fraction (HFpEF). The 5-year mortality for HFpEF has been reported as high as 50-65%. There are no current evidenced-based HFpEF therapies beyond diuretic control for fluid overload and standard treatments for comorbidities, making HFpEF an exemplary example of an unmet medical need of a rising societal burden and that is associated with substantial morbidity and mortality.

In HFpEF, sympathetic nervous system (SNS) hyperactivity results in decreased splanchnic capacitance causing more blood to be distributed into the central venous and arterial system. This leads to increase central venous pressure, pulmonary pressures and right/left heart pressures, which ultimately results in: congestions, diuretic resistance, acute decompensations leading to rehospitalization, dyspnea and intolerance to even mild exercise, and progressive diastolic dysfunction.

We believe that blocking of the GSN will stop SNS activity from reaching the splanchnic vessels and result in a redistribution of blood volume back into the splanchnic reservoir, which will result in reduction of central venous, pulmonary and right and left heart pressures. For patients with HFpEF we expect these changes to improve dyspnea and capacity to exercise, improve quality of life, increased diuretic responsiveness, Furthermore, the expected benefits of unloading the central venous and arterial system through GSN ablation should improve hemodynamic control and lessen the incidence and severity of acute decompensations leading to reduced re-hospitalizations and associated healthcare costs. This has the potential for significant social and healthcare impact.

Sympathetic and parasympathetic innervation is carried to the upper abdominal viscera by the GSN, lesser splanchnic nerve (LSN) and least splanchnic nerve (LTSN), which originate from the 5th to 8th, 9th to 10th, and 11th thoracic ganglia, respectively.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients ≥ 18 years of age with guideline defined HFpEF class III/IV (EF>40% on optimal medical therapy)
* History of exertion-related dyspnea in last 3 months
* No evidence of clinically significant peripheral edema/fluid overload
* Resting PCWP or PAD > 15 mmHg or > 25 mmHg during exercise
* The ability understand and provide signed informed consent

Exclusion Criteria:

* Myocardial infarction and/or percutaneous cardiac intervention within past 3 months; coronary artery bypass graft in past 3 months or current indication for coronary revascularization
* Admission for HF within the past month
* Systolic Blood Pressure (BP) < 120 mmHg or > 170 mmHg despite appropriate medical management
* Inability to perform Cardio Pulmonary Exercise Test (CPET)
* Presence of severe regurgitant or stenotic valve disease
* Atrial fibrillation with resting heart rate >100 beats/min
* Arterial oxygen saturation < 90 % on room air
* Significant hepatic impairment, defined as 3× upper limit of normal of transaminases, total bilirubin, or alkaline phosphatase
* Known pre-existing severe pulmonary hypertension
* Chronic pulmonary disease requiring home O2, hospitalization for exacerbation within 6 months before study entry, or on chronic steroids
* Life expectancy <12 months for non-cardiovascular reasons
* Women of childbearing age
* Currently requiring dialysis or estimated glomerular filtration rate < 40 mL/min/1.73m2
* Patients who have had cardiac transplantation or maybe considered for heart transplant
* Currently participating in an investigational drug or device study. Note: trials requiring extended follow-up for products that were investigational but have since become commercially available are not considered to be investigational trials
* Chronic or parenteral anticoagulation drug use without ability to hold for at least 72 hours
* In the opinion of the investigator, the subject is not an appropriate candidate for the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 8 (Actual)
Dates: Start 2016-08-01 (Actual); Primary Completion 2019-06-30 (Actual); Study Completion 2019-06-30 (Actual)

PRIMARY OUTCOMES:
Blunting or delay in rise of Pulmonary Capillary Wedge Pressure (PWCP) or Pulmonary Artery Diastolic Pressure (PAD) during exercise | at 1 month post-procedure as compared to baseline

SECONDARY OUTCOMES:
Reduction in resting Pulmonary Capillary Wedge Pressure (PWCP) or Pulmonary Artery Diastolic Pressure (PAD) | at 1 and 3 months post-procedure

CONTACTS AND LOCATIONS:
Locations (2):
- Na Homolce Hospital, Prague, Czechia
- 4th Military Hospital with Polyclinic, Wroclaw, Poland

IPD SHARING:
Plan to Share IPD: Undecided